CLINICAL TRIAL: NCT02937402
Title: Predictors of Response to Immune Checkpoint Inhibitors in Non-small Cell and Small Cell Lung Cancer
Brief Title: Bronchoscopy With Bronchoalveolar Lavage in Identifying Biomarkers of Response to Immune Checkpoint Inhibitors in Patients With Non-small Cell or Small Cell Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Fabien Maldonado, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC THO 16108; NCI-2016-01469 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Non-Small Cell Lung Carcinoma; Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchoscopy with bronchoalveolar lavage (Experimental): Patients undergo bronchoscopy with bronchoalveolar lavage over 45 minutes
  Interventions: Procedure: Bronchoscopy with Bronchoalveolar Lavage; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Bronchoscopy with Bronchoalveolar Lavage — Undergo bronchoscopy with bronchoalveolar lavage
Other: Laboratory Biomarker Analysis — Laboratory Biomarker Analysis

SUMMARY:
This pilot clinical trial studies how well bronchoscopy with bronchoalveolar lavage works in identifying biomarkers of response to immune checkpoint inhibitors in patients with non-small cell or small cell lung cancer. Bronchoscopy uses a thin, tube-like instrument inserted through the nose or mouth to view the inside of the trachea, air passages, and lungs. Bronchoalveolar lavage washes out the bronchi and alveoli by flushing with a fluid. Bronchoscopy with bronchoalveolar lavage may make it easier to help determine biomarkers that are more present in some cancers than others that will help determine which individuals have a greater or lesser chance of benefiting from immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To discover predictive immune biomarkers of response to immune checkpoint inhibitor therapy in individuals with primary lung cancer.

SECONDARY OBJECTIVES:

I. To determine biomarkers that may be predictive of treatment related adverse events, specifically pneumonitis.

II. To further elucidate lung immunologic microenvironment by performing single cell analysis in addition to mass cytometry (Cytof) on cells of bronchoalveolar lavage.

OUTLINE:

Patients undergo bronchoscopy with bronchoalveolar lavage over 45 minutes.

After completion of study, patients are followed up at 3, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of non-small cell lung cancer (NSCLC) or small cell lung cancer (SCLC)
* Candidate to undergo immune checkpoint inhibitor (ICI) therapy for SCLC or NSCLC (ICI as any line of chemotherapy is acceptable) as deemed by individual's treating oncologist
* Enrollment into this study may occur in tandem with other clinical therapeutics trials occurring at Vanderbilt University Medical Center (VUMC) as long as this trial does not violate protocol or inclusion criteria of that study

Exclusion Criteria:

* Coagulopathy with international normalized ratio (INR) > 2.0 or
* Coagulopathy with platelets (Plt) < 10 k
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Subjects with an active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids/immunosuppressive medications
* Respiratory failure requiring greater than 6 Lpm supplemental oxygen (O2) by nasal cannula or mechanical ventilation within the past six weeks
* Inability to perform informed consent due to any medical or psychiatric condition

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Biomarker response to immune checkpoint inhibitor therapy as measured by Response Evaluation Criteria in Solid Tumors version 1.1 criteria | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Maldonado, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided